CLINICAL TRIAL: NCT04048694
Title: Comparative Study of Calculating the Dose to the Skin by the Dosemap® Software and Its Measurement in Vivo by Gafchromic Movie
Brief Title: Comparative Study of Calculating the X-ray Dose to the Skin of the Patient Exposed
Acronym: DOSEMAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DOSEMAP
Record Dates: First submitted 2016-09-08; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Measure of the X-ray Dose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective is to estimate the precision of the calculation by the software DoseMap ® towards the in vivo measure by gafchromic movie.

DETAILED DESCRIPTION:
The procedures of Interventional Cardiology are realized under exposure in the X-rays which can be sometimes important for the patient according to the nature of the procedure.

The estimation of the dose in the skin following a procedure of interventional cardiology is difficult. The knowledge of this dose allows to anticipate the appearance of determinist effects, and so to activate a dermatological follow-up of the exposed patient in case of overtaking of a dose threshold. Unfortunately, it is impossible to measure it directly and the thresholds of exposures are fixed from the measure of the kerma in the air accumulated at the exit of the tube with X-ray, what remains very indistinct.

Since a few years the manufacturers propose tools allowing an estimation of the dose the skin of the patient. The DoseMap software ® allows to consider this dose from the data of exposure supplied by the system. To do it, it uses a modelling simplified of the patient to feign the deposit of dose in the latter.

It seems to us interesting to verify the precision of this simulation by comparing it with a measure of the in vivo dose.

ELIGIBILITY:
Inclusion Criteria:

* Procedure of Interventional Cardiology potentially more irradiant (angioplasty of the circumflex artery , or of several vessels)
* Body mass index > 25
* Collection of the Non-opposition of the patient

Exclusion Criteria:

* Diagnostic coronarography,
* Emergency procedures,
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a Interventional Cardiology procedure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Difference between the calculation by the software and the measurement by the dosimetry film | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Bourhis, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France